CLINICAL TRIAL: NCT01495572
Title: Phase II Study in Patients With Metastatic Melanoma Using a Non-Myeloablative Lymphocyte Depleting Regimen of Chemotherapy Followed by Infusion of MART-1 Reactive Peripheral Blood Lymphocytes (PBL) With or Without High Dose Aldesleukin
Brief Title: Melanoma Treatment With White Blood Cells That Destroy MART Expressing Tumor Cells
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual, the investigator decided to close the study.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Udai Kammula, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120045; 12-C-0045
Record Dates: First submitted 2011-12-16; First posted 2011-12-20 (Estimated); Results first posted 2014-06-10 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Melanoma; Skin Cancer
Keywords: Malignant Melanoma; Immunotherapy; Cell Therapy; HLA-A2 Positive; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — fludarabine; Cyclophosphamide; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Dose (HD) Aldesleukin (Experimental): Pts receiving high dose aldesleukin: Cyclophosphamide 60 mg/kg intravenous (IV) for days -7 and -6, Fludarabine 25 mg/m^2 IV for days -5 to -1, plus melanoma antigen recognized by T cells (MART)-127-35 reactive CD8+ peripheral blood lymphocytes (PBL) up to 3x10^11 IV over 20-30 minutes on day 0, plus aldesleukin 720,000 IU/kg IV over 15 minutes, every 8 hrs for up to 5 days.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Aldesleukin; Drug: MART-1 Reactive CD8+ PBL
- Peripheral Blood Lymphocytes (PBL) (Experimental): Cyclophosphamide 60 mg/kg intravenous (IV ) for days -7 and -6, Fludarabine 25 mg/m^2 IV for days -5 to -1, plus MART-127-35 reactive CD8+ PBL up to 3x10^11 IV over 20-30 minutes on day 0
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: MART-1 Reactive CD8+ PBL

INTERVENTIONS:
Drug: Fludarabine — 25 mg/m^2 IV (in the vein) for 5 days (day -5 to -1)
Drug: Cyclophosphamide — 60 mg/kg IV (in the vein) for days -7 and -6
Drug: Aldesleukin — Only given to patients assigned to high dose (HD) Arm - 720,000 IU/kg intravenous (IV) over 15 minutes, every 8 hrs (+/- 1 hr) for up to 5 days (max 15 doses).-6
  Arms: High Dose (HD) Aldesleukin
Drug: MART-1 Reactive CD8+ PBL — Intravenous (IV) over 30 minutes on day 0

SUMMARY:
Background:

- Some cancer treatments collect a patient s own blood cells to use as specialized cancer-fighting cells. Collected white blood cells known as PBL (peripheral blood lymphocytes) can use to isolate special cells that can fight tumors. Before treatment with PBL, chemotherapy is given to destroy existing white blood cells so that the new cells can survive and attack the tumors. After PBL treatment, aldesleukin is given to help the new cells grow. Researchers want to see if special white blood cells that recognize a specific protein that is present in melanoma cells (melanoma antigen recognized by T cells (MART)) can cause tumors to shrink. These white blood cells will be tested with and without aldesleukin.

Objectives:

* To test the safety and effectiveness of white blood cells that target MART in the treatment of melanoma.
* To test white blood cells that target MART with and without aldesleukin.

Eligibility:

- Individuals at least 18 years of age who have melanoma that has not responded to standard treatments.

Design:

* Participants will be screened with a medical history and physical exam. Blood and urine samples will be taken. Imaging studies such as x-rays or magnetic resonance imaging scans will be performed.
* Participants will provide white blood cells through leukapheresis. Researchers will attempt to isolate white blood cells that recognize MART
* Seven days before the start of treatment, participants will have chemotherapy.
* After the last dose of chemotherapy, participants will receive the MART reactive PBL cells. Filgrastim doses will also be given to help white blood cell counts return to normal. Participants will have frequent blood tests.
* Participants who are able to have aldesleukin treatment will start within 24 hours after receiving the MART reactive PBL cells. Treatment will continue for up to 5 days.
* Participants may have an optional tumor or lymph node biopsy to study the effects of treatment.
* If the tumor continues to grow after MART PBL treatment, participants may have one more round of cell collection and treatment.
* Participants will have followup visits for up to 6 months after receiving the MART reactive PBL treatment.

DETAILED DESCRIPTION:
Background:

* TIL transfer studies in patients with metastatic melanoma following lymphodepletion have resulted in 50 percent objective response rates with a 10-15 percent rate of complete responses. Despite these important clinical findings, adoptive cell transfer has not become widely available for patient treatment. Significant obstacles to this therapy are the need for invasive surgery and the inability of some patients to tolerate high dose aldesleukin. Further, the specific characteristics of the T cells that are responsible for the therapeutic effect of tumor infiltrating lymphocyte (TIL) are unknown, thus, resulting in significant treatment variability.
* Pre-clinical and correlative clinical studies of adoptive immunotherapy have suggested putative favorable characteristics for transferred lymphocytes, such as, high avidity for the target antigen, limited in vitro stimulation, and high expression of CD27+. However, these characteristics have not been prospectively evaluated in human clinical trials.
* We have developed a novel non invasive T cell isolation strategy using the heteroclitic MART-1:26-35(27L) peptide for in vitro sensitization of human PBL and high throughput quantitative polymerase chain reaction (qPCR) screening to rapidly isolate antigen specific cluster of differentiation 8 (CD8) + T cells from the cluster of differentiation 4 (CD4) + T cell depleted peripheral blood repertoire. These isolated T cells possess the above mentioned favorable characteristics and recognize the native MART-1:27-35 epitope, an abundantly expressed melanoma antigen presented by human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2) on the tumor surface.
* The current proposed transfer of these select MART-1:27-35 reactive lymphocytes in conjunction with a lymphodepleting preparative regimen with or without high dose aldesleukin would represent a novel therapeutic option for patients with advanced melanoma and provide a desperately needed option for patients who are not medically eligible for aldesleukin treatment.

Objectives:

* To determine whether MART-1:27-35 reactive lymphocytes infused with or without the administration of high-dose aldesleukin may result in clinical tumor regression in patients with metastatic melanoma receiving a non-myeloablative lymphoid depleting preparative regimen.
* To evaluate the safety of the treatment in patients receiving the non-myeloablative conditioning regimen and cell transfer with or without the administration of high-dose aldesleukin
* To determine the survival in patients, of infused cells following the administration of the non-myeloablative regimen, using analysis of the sequence of the variable region of the T cell receptor or flow cytometry (fluorescence activated cell sorting (FACS)).

Eligibility:

-Patients with refractory metastatic melanoma who are greater than or equal to 18 years of age, are HLA-A2+, who have MART-1:27-35 reactive peripheral blood lymphocytes available and are physically able to tolerate non-myeloablative chemotherapy. Patients must be refractory to prior high dose aldesleukin treatment if they are medically eligible to receive it. Patients who can tolerate high-dose aldesleukin will receive it with cell infusion; those who cannot tolerate high-dose aldesleukin due to medical comorbidities or refuse high-dose aldesleukin will receive cell infusion without aldesleukin.

Design:

* Patients will receive a non-myeloablative lymphocyte depleting preparative regimen consisting of cyclophosphamide (60 mg/kg/day X 2 days intravenous (IV)), fludarabine (25 mg/m^2/day IV X 5 days).
* Patients will receive intravenous adoptive transfer of MART-1:27-35 reactive peripheral blood lymphocytes (minimum 1 X 10^8 and up to a maximum of 3 X 10^11 lymphocytes) followed by high-dose intravenous (IV) aldesleukin (720,000 IU/kg/dose every 8 hours for up to 15 doses) or no aldesleukin if they are not medically eligible to receive it.
* A complete evaluation of evaluable lesions will be conducted 4-6 weeks after the last dose of aldesleukin in the aldesleukin arm and 4-6 weeks after the cell administration in the no aldesleukin arm. Patients will be enrolled into two cohorts. The cohort receiving high-dose aldesleukin will be conducted using a small optimal two-stage Phase II design, initially 19 patients will be enrolled, and if 4 or more of the first 19 patients have a clinical response ((partial response ) PR or (complete response) CR), accrual will continue to 33 patients, targeting a 35 percent goal for objective response. For the cohort who will not receive aldesleukin, the study will be conducted as a Minimax two stage phase II trial. Initially 12 evaluable patients will be enrolled to this cohort, and if 1 or more the first 12 have a response, then accrual would continue until a total of 21 patients, targeting a 20 percent goal for objective response.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable metastatic melanoma.
2. Confirmation of diagnosis of metastatic melanoma and positivity for melanoma antigens recognized by T cells (MART) confirmed by the Laboratory of Pathology of the National Cancer Institute (NCI).
3. Patients with 3 or less brain metastases are eligible. Note: If lesions are symptomatic or greater than or equal to 1 cm each, these lesions must have been treated and stable for 3 months for the patient to be eligible.
4. Patients must be refractory to high dose aldesleukin treatment.

   NOTE: This is not required for patients with non-cutaneous melanoma, patients for whom high dose aldesleukin is medically contraindicated or for patients who are unwilling to receive high dose aldesleukin.
5. MART-1:27-35 reactive peripheral blood lymphocytes derived from a leukapheresis.
6. Human leukocyte antigens (HLA-A) 0201 positive.
7. Greater than or equal to 18 years of age and less than or equal to age 70.
8. Both genders must be willing to practice birth control during treatment and for four months after receiving the preparative regimen.
9. Life expectancy of greater than three months.
10. Willing to sign a durable power of attorney.
11. Able to understand and sign the Informed Consent Document.
12. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1 for the high-dose aldesleukin cohort or ECOG 0, 1 or 2 for no aldesleukin cohort.
13. Hematology:

    * Absolute neutrophil count greater than 1000/mm^3 without support of filgrastim
    * Normal white blood cell (WBC) (> 3000/mm^3).
    * Hemoglobin greater than 8.0 g/dl
    * Platelet count greater than 100,000/mm^3.
14. Serology:

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B or hepatitis C. If hepatitis C antibody test is positive, the patients must be tested for the presence of antigen by reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative
15. Chemistry:

    * Serum alanine aminotransaminase (ALT)/aspartate aminotransaminase (AST) less than less or equal to 3 times the upper limit of normal.
    * Serum creatinine less than or equal to 1.6 mg/dl.
    * Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert s Syndrome who must have a total bilirubin less than 3 mg/dl.
16. More than four weeks must have elapsed since any prior systemic therapy, including chemotherapy, immunotherapy, and/or other targeted therapies, at the time the patient receives the preparative regimen, and patients toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients may have undergone minor surgical procedures within the past 3 weeks, as long as patients meet eligibility criteria
17. Six weeks must have elapsed from the time of any antibody therapy that could affect an anti cancer immune response, including anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) antibody therapy, so at the time the patient receives the preparative regimen to allow antibody levels to decline.
18. Patients who have previously received ipilimumab and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

NOTE: this is only required for patients who will receive high dose aldesleukin.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Systemic steroid therapy required.
3. Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
5. Opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. The following patients will be excluded from the high-dose aldesleukin arm (but may be eligible for cells alone arm):

   1. History of coronary revascularization or ischemic symptoms
   2. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45 percent.
   3. Documented LVEF of less than or equal to 45 percent tested in patients with:

      * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
      * Age greater than or equal to 60 years old
   4. Documented forced expiratory volume in 1 second (FEV1) less than or equal to 60 percent predicted tested in patients with:

      * A prolonged history of cigarette smoking (20 pk/yrs of smoking within the past 2 years)
      * Symptoms of respiratory dysfunction
   5. Clinically significant patient history which in the judgment of the Principal Investigator would compromise the patients ability to tolerate aldesleukin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udai S Kammula, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Gogas HJ, Kirkwood JM, Sondak VK. Chemotherapy for metastatic melanoma: time for a change? Cancer. 2007 Feb 1;109(3):455-64. doi: 10.1002/cncr.22427. PMID 17200963
- [Background] Rosenberg SA, Restifo NP, Yang JC, Morgan RA, Dudley ME. Adoptive cell transfer: a clinical path to effective cancer immunotherapy. Nat Rev Cancer. 2008 Apr;8(4):299-308. doi: 10.1038/nrc2355. PMID 18354418
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0045.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to slow accrual, the investigator decided to close the study.
Groups:
- High Dose (HD) Aldesleukin: Pts receiving high dose aldesleukin: Cyclophosphamide 60 mg/kg intravenous (IV) for days -7 and -6, Fludarabine 25 mg/m^2 IV for days -5 to -1, plus melanoma antigen recognized by T cells (MART)-127-35 reactive CD8+ peripheral blood lymphocytes (PBL) up to 3x10^11 IV over 20-30 minutes on day 0, plus aldesleukin 720,000 IU/kg IV over 15 minutes, every 8 hrs for up to 5 days.
  Fludarabine: 25 mg/m^2 IV (in the vein) for 5 days (day -5 to -1)
  Cyclophosphamide: 60 mg/kg IV (in the vein) for days -7 and -6
  Aldesleukin: Only given to patients assigned to high dose (HD) Arm - 720,000 IU/kg IV over 15 minutes, every 8 hrs (+/- 1 hr) for up to 5 days (max 15 doses).-6
  MART-1 Reactive CD8+ PBL: IV over 30 minutes on day 0
- Peripheral Blood Lymphocytes (PBL): Cyclophosphamide 60 mg/kg intravenous (IV ) for days -7 and -6, Fludarabine 25 mg/m^2 IV for days -5 to -1, plus MART-127-35 reactive CD8+ PBL up to 3x10^11 IV over 20-30 minutes on day 0
  Fludarabine: 25 mg/m^2 IV (in the vein) for 5 days (day -5 to -1)
  Cyclophosphamide: 60 mg/kg IV (in the vein) for days -7 and -6
  MART-1 Reactive CD8+ PBL: IV over 30 minutes on day 0
Period: Overall Study
Arm/Group | High Dose (HD) Aldesleukin | Peripheral Blood Lymphocytes (PBL)
Started | 0 | 5
Completed | 0 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High Dose (HD) Aldesleukin: Pts receiving high dose aldesleukin: Cyclophosphamide 60 mg/kg intravenous (IV) for days -7 and -6, Fludarabine 25 mg/m^2 IV for days -5 to -1, plus melanoma antigen recognized by T cells (MART)-127-35 reactive CD8+ peripheral blood lymphocytes (PBL) up to 3x1011 IV over 20-30 minutes on day 0, plus aldesleukin 720,000 IU/kg IV over 15 minutes, every 8 hrs for up to 5 days.
  Fludarabine: 25 mg/m^2 IV (in the vein) for 5 days (day -5 to -1)
  Cyclophosphamide: 60 mg/kg IV (in the vein) for days -7 and -6
  Aldesleukin: Only given to patients assigned to high dose (HD) Arm - 720,000 IU/kg IV over 15 minutes, every 8 hrs (+/- 1 hr) for up to 5 days (max 15 doses).-6
  MART-1 Reactive CD8+ PBL: IV over 30 minutes on day 0
- Peripheral Blood Lymphocytes (PBL): Cyclophosphamide 60 mg/kg intravenous (IV ) for days -7 and -6, Fludarabine 25 mg/m^2 IV for days -5 to -1, plus MART-127-35 reactive CD8+ PBL up to 3x10^11 IV over 20-30 minutes on day 0
  Fludarabine: 25 mg/m^2 IV (in the vein) for 5 days(day -5 to -1)
  Cyclophosphamide: 60 mg/kg IV (in the vein) for days -7 and -6
  MART-1 Reactive CD8+ PBL: IV over 30 minutes on day 0
- Total: Total of all reporting groups
Arm/Group | High Dose (HD) Aldesleukin | Peripheral Blood Lymphocytes (PBL) | Total
Number analyzed (Participants) | 0 | 5 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] |  | 48.4 (10.89) | 48.4 (10.89)
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 4 | 4
  >=65 years |  | 1 | 1
Gender [Number; unit: participants]
  Female |  | 2 | 2
  Male |  | 3 | 3
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native |  | 0 | 0
  Asian |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American |  | 0 | 0
  White |  | 5 | 5
  More than one race |  | 0 | 0
  Unknown or Not Reported |  | 0 | 0
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino |  | 0 | 0
  Not Hispanic or Latino |  | 5 | 5
  Unknown or Not Reported |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Tumor Response
Description: Complete response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. Partial response (PR) is at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. Progressive disease (PD) is at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study) or the appearance of one or more new lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum diameters while on study.
Time Frame: One year
Measure: Number; unit: participants
Arm/Group | High Dose (HD) Aldesleukin | Peripheral Blood Lymphocytes (PBL)
Number analyzed (Participants) | 0 | 5
participants
  Complete Response |  | 0
  Partial Response |  | 0
  Progressive Disease |  | 5
  Stable Disease |  | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events, see the adverse event module.
Time Frame: 10 months
Measure: Number; unit: participants
Groups:
- Peripheral Blood Lymphocytes (PBL): Cyclophosphamide 60 mg/kg intravenous (IV ) for days -7 and -6, Fludarabine 25 mg/m^2 IV for days -5 to -1, plus MART-127-35 reactive CD8+ PBL up to 3x1011 IV over 20-30 minutes on day 0
  Fludarabine: 25 mg/m2 IV (in the vein) for 5 days(day -5 to -1)
  Cyclophosphamide: 60 mg/kg IV (in the vein) for days -7 and -6
  MART-1 Reactive CD8+ PBL: IV over 30 minutes on day 0
Arm/Group | High Dose (HD) Aldesleukin | Peripheral Blood Lymphocytes (PBL)
Number analyzed (Participants) | 0 | 5
participants |  | 5

ADVERSE EVENTS:
Arm/Group | High Dose (HD) Aldesleukin | Peripheral Blood Lymphocytes (PBL)
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/5
Other Adverse Events (participants affected / at risk) | 0/0 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (HD) Aldesleukin (N=0) | Peripheral Blood Lymphocytes (PBL) (N=5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (HD) Aldesleukin (N=0) | Peripheral Blood Lymphocytes (PBL) (N=5)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 5 (5)
Neutrophil count decreased (Investigations) | 0 (0) | 5 (5)
Platelet count decreased (Investigations) | 0 (0) | 5 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 5 (5)

LIMITATIONS AND CAVEATS:
Due to slow accrual, the investigator decided to close the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No